CLINICAL TRIAL: NCT00414063
Title: Investigation of Differences in Energy Metabolism and Nutrient Absorption Between Lean and Obese Individuals
Brief Title: Energy Metabolism and Nutrient Absorption in Lean and Obese Individuals
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999907048; 07-DK-N048
Record Dates: First submitted 2006-12-20; First posted 2006-12-21 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2013-03-19

CONDITIONS: Obesity
Keywords: Fecal Energy; Urine Energy; Bomb Calorimetry; Gut Maintenance Flora; Obesity; Energy Metabolism
MeSH Terms: conditions — Obesity

SUMMARY:
This study will examine whether there are differences in energy (calories) losses in stool and urine between lean and obese people. People gain weight when the amount of calories in the food they eat is greater than the amount of calories their body uses to support its functions and activities. The balance between caloric intake and expenditure may be affected by the amount of calories from food that is not absorbed but is lost in stool and urine. This study will examine whether differences in food absorption are related to obesity.

Healthy normal volunteers between 18 and 45 years of age with a body mass index (BMI) of 18-25 kg/m2 or less than 35 kg/m2 may be eligible for this 15-day study. Participants are admitted to the Clinical Research Unit at the Phoenix Indian Medical Center for the study.

Participants undergo the following tests and procedures:

* Experimental diets with dye marker: Subjects are fed a 2400-calorie diet and a 3400-calorie diet for 3 days each. On the first of the day of each diet, a blue dye marker is added to the breakfast meal. A red marker is added to the breakfast meal of the first day after the diet period. Urine is collected beginning after breakfast on the first day of the diet and until before breakfast on the last day of the diet. Stool samples are collected during the entire diet period, and until the appearance of the red dye in the stool.
* 24-hour metabolic rate in the respiratory chamber: After the first diet period, subjects spend 24 hours in a respiratory chamber to measure the number of calories the body burns a day and to assess the energy balance between intake and expenditure.
* Stool sample: Stool samples are collected on days 1 and 2 of the study to look for parasites or internal bleeding that may affect nutrient absorption.
* DXA scanning: This scan uses a low dose of X-rays to measure body fat.
* Oral glucose tolerance test: For this test for diabetes, an I.V. line (needle attached to a small plastic tube) is inserted into an arm vein. The subject drinks a sugar solution. Small blood samples are drawn from the I.V. before the subject drinks the solution and at five intervals during the 3 (Omega)-hour test period.
* Fasting blood tests: On the first day of each diet and on the day after each diet is completed a blood sample is drawn before breakfast to measure hormones that may affect the ability to absorb food.

At the end of the study, some participants may be asked to repeat the experimental diets and stool and urine collections.

...

DETAILED DESCRIPTION:
The prevalence of obesity has risen to epidemic proportions in the world, resulting from both excessive energy intake and low levels of energy expenditure. The effect of nutrient absorption on energy balance, that is, the relative amount of nutrients consumed vs. the amount excreted in stool, has been reported only in small studies in which energy waste in feces and urine between lean and obese individuals was not found to be different. However, these studies were limited by small sample sizes and were not specifically designed to examine whether stool energy loss varied between lean and obese individuals. In addition, little is known about the reproducibility of the measurements of energy loss in stool and urine. We propose to investigate (i) whether there are significant differences in energy loss (as measured in stool and urine) between obese and lean individuals, and (ii) to examine the reproducibility of these measurements. Because the literature suggests a role for enteric bacterial flora in obesity, we will also examine differences in such flora between these groups. We plan to study 25 obese and 25 lean healthy non-smoking Caucasian men age 18 - 45 years old, not taking any medications (including medications for weight loss, antibiotics or probiotics) for the examination of differences in nutrient energy loss. Of these subjects, 10 lean and 10 obese individuals will be invited to repeat the study to test the reproducibility of these measurements. All participants will be admitted to the Clinical Research Unit for 15 days. During their stay, subjects will be fed a weight maintaining diet for 3 days, followed in a random cross-over design by two experimental diets: a 2400 kcal/d or 3400 kcal/d diet for 3 days. Twenty four-hour urine and feces collections will take place each day of the experimental diet period. The energy content of these waste products as well as that of the diet (using duplicate plate analysis) will be measured by bomb calorimetry. Bacterial components in feces will be extracted by repeated fractional centrifugation to obtain bacterial mass and by using 16S rDNA-based oligonucleotide probes to obtain bacterial flora. Primary results will examine the differences in energy loss between lean and obese individuals as well as the reproducibility of the measurements of stool and urine energy content.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Free of acute and chronic diseases (especially GI disorders) as determined by medical history, physical examination and laboratory tests.
* Individuals may be taking antacids and/or laxative drugs but they must be discontinued 3 or more weeks before admission.
* Age 18-45 years (in order to minimize the effect of aging on nutrient absorption).
* BMI 18-25 kg/m(2) or greater than 35 kg/m(2).

EXCLUSION CRITERIA:

* History or clinical manifestation of:

  1. Current smoking
  2. Type 2 diabetes (according to the World Health Organization diagnostic criteria)
  3. Endocrine disorders, such as Cushing's disease, pituitary disorders, and hypo- and hyperthyroidism
  4. HIV infection (self-report), due to effects on weight and body composition of HIV and medications used to treat HIV
  5. Active tuberculosis (self-report)
  6. Pulmonary disorders, including physician diagnosed chronic obstructive pulmonary diseases and obstructive sleep apnea syndrome; only subjects with mild or exercise-induced asthma on no medications or on beta-adrenergic agonists only (such as albuterol) will be allowed to enter the study
  7. Cardiovascular diseases, including coronary heart disease, heart failure, arrhythmias, and peripheral artery disease
  8. Hypertension (according to the World Health Organization diagnostic criteria), treated or uncontrolled
  9. Gastrointestinal disease, including inflammatory bowel diseases (e.g. Crohn's disease and ulcerative colitis), malabsorption syndromes (e.g. celiac disease), gastric ulcer (active)
  10. Lactose intolerance
  11. Liver disease, including non-alcoholic fatty liver disease, AST or ALT greater than 1.5 x normal value, cirrhosis, active hepatitis B or C
  12. Renal disease, as defined by serum creatinine concentrations greater than 1.5 mg/dl and/or overt proteinuria
  13. Central nervous system disease, including previous history of cerebrovascular accidents, dementia, and neurodegenerative disorders
  14. Cancer requiring treatment in the past five years, except for non-melanoma skin cancers or cancers that have clearly been cured or, in the opinion of the investigator, carry an excellent prognosis
* Behavioral or psychiatric conditions that would be incompatible with a safe and successful participation in the study (such as major depression, schizophrenia and presence of psychotic symptoms)
* Taking weight loss drugs
* Use of any antibiotic or probiotic agents within the 2 months prior to the study
* Evidence of alcohol and/or drug abuse (more than 3 drinks per day and use of drugs, such as amphetamines, cocaine, heroin, or marijuana)

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2006-12-15; Study Completion 2013-03-19

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Krakoff, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- NIDDK, Phoenix, Phoenix, Arizona, United States

REFERENCES:
- [Background] Segal KR, Dunaif A. Resting metabolic rate and postprandial thermogenesis in polycystic ovarian syndrome. Int J Obes. 1990 Jul;14(7):559-67. PMID 2228390
- [Background] Vansant G, Van Gaal L, De Leeuw I. Impact of obesity on resting metabolic rate and glucose-induced thermogenesis in non-insulin dependent diabetes mellitus. Int J Obes Relat Metab Disord. 1992 Oct;16(10):817-23. PMID 1330961
- [Background] Gougeon R, Pencharz PB, Marliss EB. Effect of NIDDM on the kinetics of whole-body protein metabolism. Diabetes. 1994 Feb;43(2):318-28. doi: 10.2337/diab.43.2.318. PMID 8288057
- [Derived] Basolo A, Parrington S, Ando T, Hollstein T, Piaggi P, Krakoff J. Procedures for Measuring Excreted and Ingested Calories to Assess Nutrient Absorption Using Bomb Calorimetry. Obesity (Silver Spring). 2020 Dec;28(12):2315-2322. doi: 10.1002/oby.22965. Epub 2020 Oct 7. PMID 33029899
- [Derived] Jumpertz R, Le DS, Turnbaugh PJ, Trinidad C, Bogardus C, Gordon JI, Krakoff J. Energy-balance studies reveal associations between gut microbes, caloric load, and nutrient absorption in humans. Am J Clin Nutr. 2011 Jul;94(1):58-65. doi: 10.3945/ajcn.110.010132. Epub 2011 May 4. PMID 21543530